CLINICAL TRIAL: NCT07119840
Title: Comparison Of Clinical Effects Of Listerine And Chlorhexidine Mouth Wash In Patients Undergoing Fixed Orthodontic Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Collaborators: Saidu College of Dentistry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMU/DIR/CTU/2025/005
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Gingivitis; Dental Plaque
Keywords: Listerine; Chlorhexidine; Gingival Index; Plaque Index; Oral Hygiene; Orthodontic Appliances
MeSH Terms: conditions — Gingivitis; Dental Plaque

STUDY DESIGN:
Intervention Model Description: A two-arm, parallel group design where participants are randomly assigned to receive either Chlorhexidine or Listerine mouthwash for 4 weeks. Each participant remains in their assigned intervention group throughout the study without crossover.
Who Masked: Participant, Care Provider
Masking Description: Participants will be randomly assigned to either the Chlorhexidine or Listerine group using a block randomization method. To ensure blinding, both mouthwashes will be dispensed in identical, unlabelled bottles. Neither the participants, the care providers will be aware of the group allocation throughout the study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Listerine Group (Experimental): Participants will receive Listerine mouthwash in unlabelled bottles once daily for 4 weeks.
  Interventions: Drug: Listerine Mouthwash Product
- Chlorhexidine Group (Active Comparator): Participants will receive chlorhexidine mouthwash in unlabelled bottles once daily for 4 weeks.
  Interventions: Drug: Chlorhexidine mouthwash

INTERVENTIONS:
Drug: Listerine Mouthwash Product — Participants in this group will receive Listerine mouthwash containing essential oils (menthol, thymol, eucalyptol, and methyl salicylate). They will be instructed to rinse once daily with 10 ml of the solution for 30 seconds after brushing, over a period of 4 weeks. The mouthwash will be dispensed in unlabelled bottles to maintain blinding. Standard oral hygiene instructions will be given.
  Other Names: Essential Oil Mouthwash
  Arms: Listerine Group
Drug: Chlorhexidine mouthwash — Participants in this group will receive Chlorhexidine mouthwash at a concentration of 0.12%. They will be instructed to rinse once daily with 10 ml of the solution for 30 seconds after brushing, over a period of 4 weeks. The mouthwash will be dispensed in unlabelled bottles to maintain blinding. Standard oral hygiene instructions will be given.
  Other Names: CHX Mouthwash
  Arms: Chlorhexidine Group

SUMMARY:
This randomized clinical trial aims to compare the effectiveness of Listerine and Chlorhexidine mouthwashes in improving periodontal health in patients undergoing fixed orthodontic treatment. Gingival Index and Plaque Index will be assessed at baseline, 2 weeks, and 4 weeks.

DETAILED DESCRIPTION:
Orthodontic treatment using fixed appliances can significantly impair oral hygiene due to the presence of brackets, bands, and wires, which create retentive areas that promote plaque accumulation. This buildup can result in gingival inflammation, leading to gingivitis or even periodontitis if not managed effectively. Mechanical plaque control, such as brushing and flossing, is often insufficient under these conditions. Thus, adjunctive chemical plaque control agents like mouthwashes are commonly recommended.

Chlorhexidine (CHX) is widely considered the gold standard for chemical plaque control due to its broad-spectrum antimicrobial activity and prolonged substantivity in the oral cavity. However, CHX is associated with side effects such as tooth staining, altered taste sensation, and mucosal irritation, limiting its long-term use. In contrast, Listerine is a commercially available essential oil-based mouthwash that has demonstrated anti-plaque and anti-inflammatory properties without the same level of side effects.

This double-blind, randomized controlled trial aims to compare the clinical efficacy of CHX (0.12%) and Listerine mouthwash in improving periodontal health among patients undergoing fixed orthodontic treatment. The study will be conducted over a period of 4 weeks at the Orthodontics Department of Saidu College of Dentistry, Swat. A total of 60 participants (30 per group), aged between 13 and 25 years, will be enrolled using non-probability consecutive sampling. Participants will be randomized into two groups using block randomization: one receiving CHX and the other Listerine, both in identical, unlabelled bottles to ensure blinding of both the investigator and participants.

The primary outcome measures are changes in Plaque Index (PI) and Gingival Index (GI), assessed at baseline (Day 0), 2 weeks, and 4 weeks. Oral examinations will be conducted by calibrated examiners using standard indices and WHO probes. Data will be analyzed using R software, with t-tests applied to compare mean scores between groups. Age and gender will be considered as potential effect modifiers.

The study is designed to evaluate whether Listerine, as a more tolerable alternative, provides comparable or superior improvements in periodontal health compared to CHX in orthodontic patients. If proven effective, Listerine may serve as a safer, more acceptable option for long-term use during orthodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 13-40 years
* Permanent dentition (including first molars)
* Willing to undergo orthodontic treatment and follow instructions

Exclusion Criteria:

* Systemic illness (e.g., diabetes, heart disease, hepatitis)
* Pregnant/lactating females
* Tobacco use
* History of allergies to mouthwash/toothpaste
* Use of mouthwash in past 3 months
* Abnormal oral morphology or parafunctional habits

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-11-29 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Gingival Index (GI) | baseline, 2 weeks, and 4 weeks , 8 week
  Measured using standard GI scale (Grades 0-3)
Plaque Index (PI) | baseline, 2 weeks, and 4 weeks , 8 week
  Measured using Orthodontic Plaque Index (Grades 0-4)

SECONDARY OUTCOMES:
Side effects | Baseline till 8 weeks
  The side effects of the trial will be noted in the adverse event log frame.

CONTACTS AND LOCATIONS:
Overall Officials: Fazli Rabi, MPH*, Principal Investigator — Khyber Medical University; Dr Naveed Sadiq, PhD, Principal Investigator — Khyber Medical University
Locations (1):
- Saidu College of Dentistry, Swāt, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No
Non Applicable

REFERENCES:
- [Background] Dehghani M, Abtahi M, Hasanzadeh N, Farahzad Z, Noori M, Noori M. Effect of Propolis mouthwash on plaque and gingival indices over fixed orthodontic patients. J Clin Exp Dent. 2019 Mar 1;11(3):e244-e249. doi: 10.4317/jced.55026. eCollection 2019 Mar. PMID 31001394
- [Background] Alavi S, Yaraghi N. The effect of fluoride varnish and chlorhexidine gel on white spots and gingival and plaque indices in fixed orthodontic patients: A placebo-controlled study. Dent Res J (Isfahan). 2018 Jul-Aug;15(4):276-282. PMID 30123305
- [Background] Priya BM, Anitha V, Shanmugam M, Ashwath B, Sylva SD, Vigneshwari SK. Efficacy of chlorhexidine and green tea mouthwashes in the management of dental plaque-induced gingivitis: A comparative clinical study. Contemp Clin Dent. 2015 Oct-Dec;6(4):505-9. doi: 10.4103/0976-237X.169845. PMID 26681856
- [Background] Zuttion GS, Juarez HAB, Lima BD, Assumpcao DP, Daneris AP, Tuchtenhagen IH, Casarin M, Muniz FWMG. Comparison of the anti-plaque and anti-gingivitis efficacy of Chlorhexidine and Malva mouthwashes: Randomized crossover clinical trial. J Dent. 2024 Nov;150:105313. doi: 10.1016/j.jdent.2024.105313. Epub 2024 Aug 22. PMID 39173823
- [Background] Atassi F, Awartani F. Oral hygiene status among orthodontic patients. J Contemp Dent Pract. 2010 Jul 1;11(4):E025-32. PMID 20953561